CLINICAL TRIAL: NCT03796923
Title: Models of Care in the Transition From the Secondary to the Primary Sector Among the Frailest Elderly +75; a Randomized Controlled Trial
Brief Title: Models of Care in the Transition From the Secondary to the Primary Sector Among the Frailest Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MOCATRANFRAELRCT
Record Dates: First submitted 2019-01-02; First posted 2019-01-08 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Frail Elderly Syndrome; Transitional Care; Frailty; Readmission; Aging; Elderly
Keywords: Elderly; Hospital at home; Readmission; Transitional care; Frailty; Patient Related Outcome Measures
MeSH Terms: conditions — Frailty | interventions — Geriatric Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention I (Active Comparator): Intervention (I): early follow-up visit from the community nurse within 24 hours after discharge
  Interventions: Other: Early follow-up visit after discharge; Other: Comprehensive geriatric assessment (CGA)
- Intervention II (Experimental): Intervention (II): early follow-up by the geriatric team within 24 hours after discharge
  Interventions: Other: Early follow-up visit after discharge; Other: Comprehensive geriatric assessment (CGA); Other: Continued geriatric care
- Control (Other): Usual care: individualized follow-up performed by the GP and municipality services
  Interventions: Other: Possible follow-up visit from GP

INTERVENTIONS:
Other: Early follow-up visit after discharge — Early follow-up visit and different degrees of specialized care after discharge
  Arms: Intervention I; Intervention II
Other: Comprehensive geriatric assessment (CGA) — Comprehensive geriatric assessment (CGA) during admission
  Arms: Intervention I; Intervention II
Other: Continued geriatric care — Continued specialized geriatric care after discharge
  Arms: Intervention II
Other: Possible follow-up visit from GP — Usual care: follow up visit from GP within one week after discharge
  Arms: Control

SUMMARY:
In most Western countries the elderly population increases rapidly. In Denmark, the population of elderly aged 75 years or older may amount to nearly 15 % of the entire population in 2050 compared to 9 % today (2017). A large part of the elderly population is at high risk of hospitalization including more admissions and increased morbidity and mortality. The number of hospital beds is declining persistently, calling for shorter lengths of stay (LOS). Increasingly complex treatments now take place outside hospital. Presently, many Danish regional hospitals establish geriatric wards and other geriatric in-hospital and outpatient services to overcome these challenges. The aim of the present PhD-study is to investigate the effects of different models of transitional care among the frailest elderly patients.

DETAILED DESCRIPTION:
Design Population: The frailest acutely admitted geriatric patients aged +75. Intervention: Early follow-up visits after discharge. Comparison: Usual care follow-up. Outcomes: The primary outcome is readmission within 30 days after discharge. Secondary outcomes are: mortality 30 days after discharge and 90 days after admission, length of stay (LOS), direct discharge from the Emergency Department, time at home before readmission, duration of readmission and physical functional status 30 days after discharge.

Methods The first study is conducted as a randomized controlled trial (RCT) using two different degrees of intervention. The second study is a cohort study of an unexposed control group. The third study is sub-group analyses of the RCT data according to frailty status and type of dwelling.

A focus group comprised of included patients and relatives will be set to identify additional patient related outcome measures (PROMs) and to participate in an advisory group throughout the remaining project.

ELIGIBILITY:
Inclusion Criteria

* Aged 75 years or older
* Living within the municipality of Aarhus (except for the control group, see below)
* MPI-score = 2 (moderate frailty) or MPI score = 3 (severe frailty)

Exclusion Criteria

* Included in any other kind of follow-up schemes
* Declared terminally ill or undergoing palliative care at admission
* Admitted from one specific temporary nursing home with geriatric medical assistance
* Discharge or transfer to another department, including hospice
* MPI-score = 1 (low frailty)
* Discharged to one specific temporary nursing home with geriatric medical assistance
* The patient does not want a visit after discharge

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 3340 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
Readmission | 30 days
  Readmission within 30 days after discharge

SECONDARY OUTCOMES:
Mortality | 90 days after admission and 30 days after primary discharge
  Mortality within 90 days after admission and 30 days after discharge
Length of stay (LOS) | 30 days after primary discharge
  Length of stay during primary admission and total length of stay including following readmissions

OTHER OUTCOMES:
Physical functional status 30 days after discharge | 30 days after discharge
  Functional Recovery Score ADL and Functional Recovery Score I-ADL: sum-score, range 100-0 (100 is the highest physical functional status score possible, 0 is the lowest)
Duration of readmission | 30 days after discharge
  Duration of readmission
Time at home before readmission | 30 days after discharge
  Time at home before readmission
Number of patients discharged directly from the Emergency Department (ED) | 30 days after discharge
  Patients discharged directly from the ED

CONTACTS AND LOCATIONS:
Overall Officials: Else Marie S Damsgaard, Prof., DMSci, Study Chair — University of Aarhus
Locations (1):
- Aarhus University, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hansen TK, Pedersen LH, Shahla S, Damsgaard EM, Bruun JM, Gregersen M. Effects of a new early municipality-based versus a geriatric team-based transitional care intervention on readmission and mortality among frail older patients - a randomised controlled trial. Arch Gerontol Geriatr. 2021 Nov-Dec;97:104511. doi: 10.1016/j.archger.2021.104511. Epub 2021 Aug 26. PMID 34479071

DOCUMENTS (1):
  • Study Protocol (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/23/NCT03796923/Prot_002.pdf